CLINICAL TRIAL: NCT04818164
Title: Prone Position Improves End-Expiratory Lung Volumes in COVID-19 Associated Acute Respiratory Distress Syndrome: An Observational Study
Brief Title: Prone Position Improves End-Expiratory Lung Volumes in COVID-19 Acute Respiratory Distress Syndrome
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Olcay Dilken, Principal Investigator, Istanbul University - Cerrahpasa
Other Study IDs: 2020-19-16163
Record Dates: First submitted 2021-03-25; First posted 2021-03-26 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-03

CONDITIONS: Acute Respiratory Distress Syndrome; Coronavirus; Mechanical Ventilation Complication; Ventilation Perfusion Mismatch
Keywords: acute respiratory distress syndrome; prone position; lung recruitment
MeSH Terms: conditions — Respiratory Distress Syndrome; Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Covid-19 associated Acute Respiratory Distress Syndrome (ARDS) may present with profound hypoxemia not fully explained with pulmonary infiltrates. Accordingly, how prone positioning improves oxygenation in these patients is not fully known. The investigators conducted a study among patients with severe Covid-19 ARDS receiving prone position for at least 16 hours. End Expiratory Lung Volume (EELV) was measured with Nitrogen wash-in/wash-out technique before (Supine Position 1- SP1), during (Prone Position - PP) and after (Supine Position 2 - SP2) prone positioning.

DETAILED DESCRIPTION:
After initiation of invasive mechanical ventilation, initial ventilator settings were performed by the attending physician. These settings include titration of best PEEP to promote oxygenation if Spo2 <92% despite a Fio2 higher than 80% or best compliance that do not jeopardize oxygenation if Fio2 is between 50-80% and Spo2 >92%. After a period of 30 minutes for stabilisation, the first set of measurements were done in the SP1 position. Afterwards, the patient was turned to prone position with the same PEEP (which was unchanged throughout the study period) and measurements were repeated every four hours until the patient was reverted back to SP2. Eventually, there were 7 measurements in total. (SP1, PP0, PP4, PP8, PP12, PP16, SP2). Dead space ventilation and shunt fraction calculations were made based on central venous blood gas measurements and oxygen consumption and carbon dioxide production at the relevant timepoint.

ELIGIBILITY:
Inclusion Criteria:

* Patients were considered eligible if they met the Berlin definition criteria for ARDS and intubated due to increased work of breathing and/or worsening hypoxemia. All patients had a positive Covid-19 real time Polymerase Chain Reaction test

Exclusion Criteria:

* Exclusion criteria were; age < 18 years, ARDS resulting from other risk factors, presence of chest drainage tubes, tracheostomy, pneumomediastinum, hemodynamic instability (systolic blood pressure < 100 mmHg, lactate > 2 mmol/l, or an increase in lactate concentrations for 20% in two consecutive blood gas analysis within 2 hours interval) and suspicion or confirmed pulmonary emboli.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Patients receiving invasive mechanic ventilation due to Covid-19 ARDS
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Partial Pressure of Oxygen/ Fraction of Inspired Oxygen | 1 day
  Oxygenation
End Expiratory Lung Volume | 1 day
  Oxygenation

SECONDARY OUTCOMES:
Lung Compliance | 1 day
  Change in Recruitable Lung Volume
Dead Space Ventilation | 1 day
  Fraction of Wasted Ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Olcay Dilken, Dr., Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpaşa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dilken O, Rezoagli E, Yartas Dumanli G, Urkmez S, Demirkiran O, Dikmen Y. Effect of prone positioning on end-expiratory lung volume, strain and oxygenation change over time in COVID-19 acute respiratory distress syndrome: A prospective physiological study. Front Med (Lausanne). 2022 Dec 2;9:1056766. doi: 10.3389/fmed.2022.1056766. eCollection 2022. PMID 36530873